CLINICAL TRIAL: NCT00402311
Title: A Prospective Randomized Trial on the Effects of a Psychogeriatric Diagnostic Day Hospital
Brief Title: The Effects and Cost-Effectiveness of an Integrated Multidisciplinary Approach for Psychogeriatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 945-02-055
Record Dates: First submitted 2006-11-20; First posted 2006-11-22 (Estimated); Last update posted 2007-01-22 (Estimated); Status verified 2006-11

CONDITIONS: Delirium, Dementia, Amnestic, Cognitive Disorders; Memory Disorders
Keywords: Health Services for the Aged; Geriatric Psychiatry
MeSH Terms: conditions — Neurocognitive Disorders; Memory Disorders

INTERVENTIONS:
Procedure: DOC-PG: integrated multidisciplinary assessment
Procedure: Usual care: assessment by GP or one of the regional services

SUMMARY:
The purpose of this study is to determine the effects and cost-effectiveness of a Diagnostic Observation Center for PsychoGeriatric patients (DOC-PG). Our main hypothesis is that DOC-PG has added value compared with usual care regarding Health Related Quality of Life (HRQoL).

DETAILED DESCRIPTION:
An integrated multidisciplinary approach to diagnosing and managing dementia is generally recommended, though rarely investigated. In recent years, multidisciplinary memory clinics (MCs) for patients with dementia have been established in many places over the world. These services have recently also been criticised for being principally hospital-based, for their apparently limited focus that entails only medical diagnostics and pharmacotherapy and for thus diverting resources from community mental health teams(CMHTs) .On the other hand, CMHTs are mainly concerned with the provision and organisation of integrated care, and unlike MCs, CMHTs generally have limited access to hospital-based diagnostics such as brain-imaging.

In April 2002, an outpatient diagnostic facility, the Diagnostic Observation Centre for PsychoGeriatric patients (DOC-PG) was established in Maastricht, the Netherlands. DOC-PG combines the hospital-based approach of the MC with the care-oriented approach of the regional CMHT and aims to provide the general practitioner (GP) with elaborate diagnostic and therapeutic advice for patients with cognitive disorders.

Comparison: DOC-PG is compared with usual care i.e. the GP took care of the diagnosis, or he or she referred the patient to one of the separate regional services, e.g. the Maastricht Memory Clinic (MMC), geriatric medicine, or the department of mental health for the elderly of the mental health community service (CMHT).

ELIGIBILITY:
Inclusion Criteria:

* Aged 55 years or over
* Suspected of having dementia or combined somatic/psychiatric disorder
* No referral to other local/regional services in the last two years
* Availability of a proxy (visiting the patient at least once a week)

Exclusion Criteria:

* Acute disorders that need a prompt therapeutic intervention
* Living in a nursing home or receiving care that is comparable to that of a nursing home

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216
Dates: Start 2002-04; Study Completion 2005-08

PRIMARY OUTCOMES:
The Visual Analogue Scale of the EuroQol-5D

SECONDARY OUTCOMES:
Utility score of the EuroQol-5D
Short Form 36 (SF-36)
Mini Mental State Examination (MMSE)
Global Deterioration Scale (GDS)
NeuroPsychiatric Inventory (NPI)
Instrumental Activities of Daily Living scale (IADL)
Cornell Scale of Depression in Dementia (CSDD)
Perceived Pressure from Informal Care (Dutch translation, EDIZ)
Informal care questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Frans R Verhey, PhD, MD, Principal Investigator — Maastricht University Medical Center; Carmen D. Dirksen, PhD, Study Director — Maastricht University Medical Center; Johan L Severens, PhD, Study Director — Maastricht University Medical Center; Alfons Kessels, MD, MSc, Study Chair — Maastricht University Medical Center; Claire A Wolfs, MSc, Study Chair — Maastricht University Medical Center
Locations (1):
- Academic Hospital Maastricht, Maastricht, Limburg, Netherlands

REFERENCES:
- [Background] Wolfs CA, Dirksen CD, Severens JL, Verhey FR. The added value of a multidisciplinary approach in diagnosing dementia: a review. Int J Geriatr Psychiatry. 2006 Mar;21(3):223-32. doi: 10.1002/gps.1454. PMID 16440403
- [Background] Wolfs CAG, Severens JL, Dirksen CD, Kessels A, Jaspers N, Verhey FRJ. 2005. A Randomized Clinical Trial on the Effects of a Diagnostic Observation Centre for PsychoGeriatric patients (DOC-PG). International Psychogeriatrics 17: 370-371
- [Result] Wolfs CA, Verhey FR, Kessels A, Winkens RA, Severens JL, Dirksen CD. GP concordance with advice for treatment following a multidisciplinary psychogeriatric assessment. Int J Geriatr Psychiatry. 2007 Mar;22(3):233-40. doi: 10.1002/gps.1666. PMID 16977677
- [Derived] Wolfs CA, Dirksen CD, Kessels A, Severens JL, Verhey FR. Economic evaluation of an integrated diagnostic approach for psychogeriatric patients: results of a randomized controlled trial. Arch Gen Psychiatry. 2009 Mar;66(3):313-23. doi: 10.1001/archgenpsychiatry.2008.544. PMID 19255381
- See also: Related Info — http://www.alzheimercentrumlimburg.nl/